CLINICAL TRIAL: NCT04112433
Title: Novel Cardiac Signal Processing System for Electrophysiology Procedures
Brief Title: Novel Cardiac Signal Processing System
Status: Completed | Type: Observational
Sponsor: BioSig Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PURE EP 2.0
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrhythmia
Keywords: Cardiac Signal; Ablation; Signal Processing; Intracardiac Electrogram; Electrophysiology; Electrogram; Signals; Cardiac; Cardiac Ablation; Atrial fibrillation; Atrial Flutter; Ventricular Tachycardia; Arrhythmias; PVC's
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bioelectrical cardiac signals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PURE EP 2 Group: Enrolled and consented patients who are indicated for and receive an elective cardiac ablation procedure using the PURE EP 2 system for monitoring and collection of intracardiac electrogram signals.
  Interventions: Device: PURE EP 2

INTERVENTIONS:
Device: PURE EP 2 — Enrolled patients receiving cardiac ablation treatment using the current standard of care with additional monitoring and intracardiac electrogram signal collection via the PURE EP 2 system.

SUMMARY:
This study is designed to collect parallel intracardiac signal data during pre-defined periods of clinical interest from the PURE EP system and the existing signal recording and mapping systems.

The collected signals will then undergo BLINDED, CONTROLLED evaluation by unbiased electrophysiologist reviewer(s) to determine whether the PURE EP signals provides additional or clearer diagnostic information.

DETAILED DESCRIPTION:
Cardiac electrophysiologists rely on the display of electrograms when performing electrophysiology (EP) studies and catheter ablations in patients with arrhythmias. To achieve effective outcomes without complications, it is vital that the recording system enables the recognition of clearly abnormal (scared myocardium) and normal electrical signals.

Current recording systems have limitations in that it can be difficult to clearly distinguish a true cardiac signal from noise or artifact. This is particularly true when pacing the heart and when ablating abnormal myocardial tissue, components of the conduction system or epicardial structures. Therefore, improvement of the fidelity of signals obtained from EP recording systems is needed to enhance identification of the most effective targets for ablation.

There are several standard electrophysiology recording systems in use today, such as the commonly used GE/Prucka CardioLab recording system ("Prucka") which would benefit from additional features in order to improve the ability to record, discriminate and analyze signals from the heart. BioSig Technologies, Inc. ("BioSig") has developed an electrophysiology signal processing system, the PURE EP™ System, which may allow electrophysiologists to better characterize arrhythmogenic tissue during ablation procedures. Specifically, the PURE EP™ System's higher sampling rate and higher dynamic range allow improved visualization of low amplitude signals, especially those temporally situated near low frequency, high amplitude signals or large high-frequency signals.

This multi-center, prospective, non-randomized, observational study will involve at least five patients undergoing elective cardiac ablation procedure for tachycardias such as atrial fibrillation, atypical atrial flutter, ischemic ventricular tachycardia, or symptomatic premature ventricular contractions (PVCs). The existing recording/mapping system clocks will be synchronized to the PURE EP clock prior to each procedure. At the beginning of the procedures, all systems will be optimized for best signal display based on the physician preference. During the ablation procedures, annotations will be captured on the PURE EP system based on pre-determined clinically relevant events defined in this protocol (example - before and after successful ablation therapy).

After the procedures, parallel signal data samples will be harvested from all the systems using the procedure annotations and the time stamps as a guide. Once the signal data is harvested, cleaned, and organized, the individual signal samples will be reviewed in a blinded, controlled fashion by a group of independent, unbiased electrophysiologist(s).

Selected signal sample sets (from the same date and time stamp) will be separated in the survey and arranged in random order. The reviewer will be asked specific and identical questions relevant to each set of signal samples, but the individual samples will be separated and randomized across a full survey containing many different signal samples from many different procedures. The signal survey will be created under the direction of the Principle Investigator. The selection of the independent EP reviewers will also be done under the direction of the Principle Investigator

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac ablation treatment
* Signed informed consent

Exclusion Criteria:

* contraindication to electrophysiology study or ablation
* Enrollment in any other ongoing arrhythmia study protocol
* Active Infection or sepsis
* Pregnancy or lactation
* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person indicated and consented for an elective cardiac ablation procedure who is >18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Safe and effective use of the PURE EP 2 system based on system specifications and recorded within the Case Report Form (CRF). | Throughout the cardiac ablation procedure
  The primary aim of this study is to further establish the safe and effective use of the PURE EP System during cardiac ablation in the EP Laboratory in a post-market environment. The PURE EP System will be installed to run in parallel to existing mapping and recording systems already in use in the EP lab. Each system will be optimized for viewing intracardiac signals based on the physician preference. The existing systems will serve as the primary method of viewing intracardiac signals and the PURE EP system will be redundant.
  The intracardiac signals from the PURE EP system will be compared to existing recording and mapping system signals generated in real-time during each ablation procedure. The PURE EP system signals will be monitored by the physician investigator and a company clinical representative to validate the PURE EP 2 system runs as intended based on the system manual and meets expected standards for displaying signals.

SECONDARY OUTCOMES:
Assess the quality of the PURE EP 2 intracardiac signals when compared to existing recording and mapping systems as determined by controlled survey of blinded, independent expert electrophysiology reviewers. | After the collection of signal samples from at least (5) subjects and until study completion
  The secondary aim of this study is to assess the quality of the PURE EP intracardiac signals and the associated clinical relevance of the signals when compared to other sources of intracardiac signals. During the ablation procedures, annotations will be captured on the PURE EP system based on clinically relevant events defined in the protocol.
  After the procedure, parallel signal data samples will be harvested from all the systems using annotations and the time stamps as a guide. Once the signal data is harvested and organized, the signal samples across multiple procedures will be reviewed in a blinded, controlled fashion by 2-3 independent, unbiased expert electrophysiologist(s).
  The sample survey will be created under the direction of the PI.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. David's Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Collected intracardiac signal samples will be shared with the independent electrophysiologist reviewers, other physician investigators, and possibly other study collaborators like a biostatistician and clinical research organization.

REFERENCES:
- [Derived] Padmanabhan D, Sugrue A, Vaidya V, Witt C, Yasin O, Naksuk N, Killu A, Foxall T, Drakulic BS, Venkatachalam KL, Asirvatham SJ. Incremental benefit of a novel signal recording system during mapping and ablation. Europace. 2021 Jan 27;23(1):130-138. doi: 10.1093/europace/euaa194. PMID 33094311